CLINICAL TRIAL: NCT00653718
Title: Musculoskeletal Pain in Postmenopausal, Early Breast Cancer Patients Receiving Aromatase Inhibitor Therapy - A Pilot Study
Acronym: AIMS
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5390L00068
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2008-09

CONDITIONS: Breast Cancer
Keywords: Pain; Characterize musculoskeletal pain; Breast cancer patients treated with aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In 2005, the EBCIG demonstrated the efficacy of tamoxifen in improving overall survival in hormone receptor positive breast cancers. However, tamoxifen shows partial estrogen agonist activity, which is responsible for the drug's detrimental effects such as endometrial carcinoma, thromboembolism, and tamoxifen resistance. More recently, aromatase inhibitors have been shown to be superior to tamoxifen in the metastatic and adjuvant settings. The ATAC trial demonstrated improved disease-free survival (DFS) for 5 years of anastrozole compared to 5 years of tamoxifen 3. The BIG 1-98 trial results demonstrated that after a median follow-up of 25.8 months, letrozole improved DFS and distant DFS when compared to tamoxifen. Based on these results, adjuvant hormonal therapy with Aromatase Inhibitors (AI) has become the preferred therapy for post-menopausal woman.

However, AI therapy is also associated with toxicities that merit in-depth studies, one of them being an increase in musculoskeletal pain. In the ATAC trial, at a median follow-up of 5.7 years, arthralgia was significantly higher (35.6% vs. 29.4%) and fractures were also increased (11.0% vs. 7.7%) when anastrozole was administered for 5 years following surgery with or without chemotherapy 3. The incidence of arthralgia was also significantly higher in the MA-17 trial, with 25% of patients receiving letrozole developing arthralgia compared with 21% in the placebo group following 5 to 6 years of tamoxifen 5.

Traditionally in cancer clinical trials, the reporting of musculoskeletal pain has been based on the "Common Terminology Criteria for Adverse Events", which covers a wide range of symptoms and does not facilitate the documentation of a pain syndrome in a specific manner. Therefore, there is a need to design a study that will describe the nature of the pain associated with the administration of AI therapy using tools that have been validated for capturing a multidimensional phenomenon such as pain.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Invasive carcinoma of the breast confirmed by needle biopsy or final pathological evaluation of the surgical specimen
* Breast cancer Stage I, II or IIIa
* ER and/or PR+
* No evidence of metastatic disease
* Post-menopausal
* May or may not have received adjuvant or neoadjuvant chemotherapy
* Bilateral infiltrating carcinoma are eligible

Exclusion Criteria:

* Men not eligible
* Other malignancies
* Patients who have received neoadjuvant or adjuvant endocrine therapy with tamoxifen or an aromatase inhibitor
* Ongoing treatment with any sex hormonal therapy (these patients are eligible if this therapy is discontinued prior to entry)
* Therapy with hormonal agent such as raloxifene for osteoporosis
* Patients receiving glucocorticoids
* Psychiatric or addictive disorders
* Inability to read English or French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal pain | Every two weeks

SECONDARY OUTCOMES:
Lymphocyte gene expression profiling | Every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: André Robidoux, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada